CLINICAL TRIAL: NCT07104370
Title: Comparison of Freeze-dried Bone Allograft and Autogenous Bone Blocks in the Surgical Reconstruction of Horizontally Atrophied Jaws for Implant Placement: Randomized Clinical Trial
Brief Title: Freeze-dried Bone Allograft vs Autologous Bone Blocks in the Lateral Augmentation of the Jaws
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Szerencse Csilla, Dentist, oral surgeon, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEDCD45
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Edentulous Alveolar Ridge; Edentulous Alveolar Ridge Atrophy
Keywords: autologous bone; retromolar area; bone block; bone augmentation; dental implant; freeze-dried bone allograft
MeSH Terms: interventions — formycin diphosphate; Bone Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Freeze-dried allograft bone block (Experimental): A freeze-dried bone allograft block is used for the lateral augmentation of the atrophied jaw.
  Interventions: Procedure: Bone augmentation using freeze-dried allograft block; Diagnostic Test: preoperative cone beam computed tomography (CBCT); Diagnostic Test: post-operative cone beam computed tomography (CBCT); Procedure: Dental implant placement; Diagnostic Test: Bone core biopsy; Procedure: Fixed dental prosthesis (FDP) fabrication; Device: Bone grafting
- Autogenous bone block (Active Comparator): An autogenous bone block harvested from the retromolar area of the mandible is used for the lateral augmentation of the atrophied jaw.
  Interventions: Procedure: Bone augmentation using an autologous bone block; Diagnostic Test: preoperative cone beam computed tomography (CBCT); Diagnostic Test: post-operative cone beam computed tomography (CBCT); Procedure: Dental implant placement; Diagnostic Test: Bone core biopsy; Procedure: Fixed dental prosthesis (FDP) fabrication

INTERVENTIONS:
Procedure: Bone augmentation using an autologous bone block — * Under local anesthesia, a crestal and mesial releasing incision is made, followed by preparation of a full-thickness mucoperiosteal flap.
  * In the control group, an autologous bone block graft is harvested from the retromolar donor area using rotary instruments and piezoelectric surgery.
  * The block is fixed to the recipient site with two screws.
  * The flap is mobilized, and the wound is closed tension-free with mattress and simple interrupted sutures.
  * Sutures are removed two weeks postoperatively.
  * All patients receive therapeutic-dose antibiotics: amoxicillin and clavulanic acid 2x1 for one week. In the case of an amoxicillin allergy, clindamycin 4x1 for seven days is administered. Non-steroid anti-inflammatory treatment with diclofenac 3x1 is also provided.
  * Patients do not wear temporary prostheses during the healing period.
  Arms: Autogenous bone block
Procedure: Bone augmentation using freeze-dried allograft block — * Under local anesthesia, a crestal and mesial releasing incision is made, followed by preparation of a full-thickness mucoperiosteal flap.
  * In the test group, a freeze-dried allograft bone block is prepared to the required size using rotary instruments.
  * The block is fixed to the recipient site with two screws.
  * The flap is mobilized, and the wound is closed tension-free with mattress and simple interrupted sutures.
  * Sutures are removed two weeks postoperatively.
  * All patients receive therapeutic-dose antibiotics: amoxicillin and clavulanic acid 2x1 for one week. In case of amoxicillin allergy, clindamycin 4x1 for seven days is administered. Non-steroid anti-inflammatory treatment with diclofenac 3x1 is also provided.
  * Patients do not wear temporary prostheses during the healing period.
  Arms: Freeze-dried allograft bone block
Diagnostic Test: preoperative cone beam computed tomography (CBCT) — • Preoperatively, a CBCT scan is performed to assess inflammatory and other pathological changes and anatomical variations in the dentomaxillofacial region.
Diagnostic Test: post-operative cone beam computed tomography (CBCT) — Postoperatively, a CBCT scan is performed to assess bone quantity and quality before implantation.
Procedure: Dental implant placement — Following the 3-month-long healing period following bone augmentation, dental implants are placed non-submerged in the augmented bone under local anaesthesia.
Diagnostic Test: Bone core biopsy — At the time of dental implant placement, a rotary instrument is used to harvest a bone core biopsy sample from the augmented bone. The bone core biopsy samples are subjected to histomorphometric and microCT analysis.
Procedure: Fixed dental prosthesis (FDP) fabrication — After 3 months of dental implant placement, fixed dental prosthesis are delivered on the dental implants.
Device: Bone grafting — Freeze-dried bone allograft block
  Arms: Freeze-dried allograft bone block

SUMMARY:
After tooth loss, the alveolar ridge undergoes various modeling and remodeling processes, resulting in overall bone resorption. In case of extensive alveolar atrophy, bone volume must be restored before or during implant placement to achieve successful dental rehabilitation and maximize implant survival and success rates. One possible method for reconstructing severe bone resorption is block bone augmentation.

Due to its biological properties, autologous bone is considered the "gold standard" among bone graft materials, as it possesses osteoinductive, osteoconductive, and osteogenic properties.

The advantages of using allografts over autologous bone grafts include reduced postoperative morbidity, decreased surgical time, and the absence of anatomical limitations regarding the amount of bone that can be harvested. The disadvantage of allografts is the loss of viable osteogenic cells and osteoinductive factors during processing.

The aim of the study is:

* to compare the success of the bone augmentation surgery depending on whether freeze-dried bone allograft blocks or autologous bone blocks are used,
* compare the microarchitecture of the augmented bone depending on the bone graft material applied,
* to evaluate the success of dental implants placed in the augmented bone and that of the prostheses delivered on the dental implants.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* require lateral augmentation for implant rehabilitation

Exclusion Criteria:

* Smoking
* Pregnancy
* Poor oral hygiene
* Failure to attend follow-up visits
* Therapeutic-dose irradiation to the head and neck region
* Local bone tumors, cysts, or inflammatory processes
* Decompensated systemic diseases contraindicate surgery
* Use of medications affecting bone metabolism (steroids, antiresorptive medications such as bisphosphonates, RANKL inhibitor antibodies, VEGF antagonists)
* Psychiatric disorders contraindicate implant rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
Success of the bone augmentation | 3 months
  The bone augmentation surgery is successful if no inflammatory complications occur in the 3-month healing period and the bone volume is sufficient for dental implant placement.
Success of the dental implants | 3 months
  According to The International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference.
  I. Success (optimum health)
  1. No pain or tenderness upon function
  2. 0 mobility
  3. Less than 2 mm radiographic bone loss from initial surgery
  4. No exudates in the patient's history
  II. Satisfactory survival
  1. No pain on function
  2. 0 mobility
  3. 2-4 mm radiographic bone loss
  4. No exudates in the patient's history
  III. Compromised survival
  1. May have sensitivity to the function
  2. No mobility
  3. Radiographic bone loss of more than 4 mm (less than1/2 of the length of the implant body)
  4. Probing depth more than 7 mm
  5. May have exudates in the patient's history
  IV. Failure (clinical or absolute failure)
  Any of the following:
  1. Pain on function
  2. Mobility
  3. Radiographic bone loss of more than 1/2 the length of the implant
  4. Uncontrolled exudate
  5. Implant no longer in the mouth
Success of the implant-borne prostheses | 5 years
  Prostheses with four or fewer complications (screw loosening, decementation, chipping) that could be treated chairside.

SECONDARY OUTCOMES:
Hisomorphometry: Percent of residual bone graft particles | 3-6 months
  The percentage of residual bone graft particle area measured on the representative sections prepared from the bone core biopsy samples. Unit: percent (%)
Hisomorphometry: Percent of newly formed bone | 3-6 months
  The percentage of newly formed bone area is measured on the representative sections prepared from the bone core biopsy samples. Unit: percent (%).
Hisomorphometry: Percent of bone marrow | 3-6 months
  The percentage of bone marrow area measured on the representative sections prepared from the bone core biopsy samples. Unit: percent (%)
Value of the percent bone volume (BV/TV) calculated from the microCT reconstructions of the bone core biopsy samples | 3-6 months
  Relative volume of calcified tissue in the selected volume. Unit: none
Value of the bone surface to volume ratio (BS/TV), calculated from the microCT reconstructions of the bone core biopsy samples | 3-6 months
  Ratio of the segmented bone surface to the total volume in the region of interest. Unit: 1/mm
Value of the trabecular thickness (Tb.Th.) calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Mean thickness of the trabeculae, assessed using direct 3D methods. Unit: mm.
Value of the trabecular separation (Tb.Sp.), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Mean distance between the trabeculae, assessed using direct 3D methods. Unit: mm.
Value of the trabecular bone pattern factor (Tb.Pf), derived from microCT reconstructions of bone core biopsy samples. | 3-6 months
  An indicator of the relation between convex and concave elements in the trabecular bone structure. Tb.Pf <0 when the trabecular bone is honeycomb-like and increases as the trabecular bone acquires a rod-like structure. Unit: none.
Value of the structure model index (SMI), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  The estimator of the plate-versus rod-like characteristic of the trabecular bone structure, 0 for perfect plates, 3 for perfect rods, and 4 for perfect spheres. Unit: none.
Value of the Total porosity (Po(tot)), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Percent porosity is the volume of pores as a percent of the total volume of interest (VOI). Unit: percent (%).
Value of the Connectivity (Conn), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  One useful and fast algorithm for calculating the Euler connectivity in 3D is the "Conneulor". It measures what might be called "redundant connectivity", the degree to which parts of the object are multiply connected. It is a measure of how many connections in a structure can be severed before the structure falls into two separate pieces. Unit: none.

CONTACTS AND LOCATIONS:
Overall Officials: Csilla Szerencse, DMD, MDS, Principal Investigator — Department of Public Dental Health Semmelweis University
Locations (1):
- Semmelweis University Department of Public Dental Health, Budapest, Hungary, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published after de-identification.
Supporting Information: Study Protocol
Time Frame: Immediately after publication, no end date
Access Criteria: Anyone who wishes access the data.